CLINICAL TRIAL: NCT06537401
Title: Adaptations in Postprandial Metabolic Flexibility Following a Three-day, High-fat Diet
Brief Title: Metabolic Adaptations to High-fat Diet
Acronym: MetFlexHFD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility of subjects completing the 3 day high fat diet protocol and multiple oral glucose tests
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Matthew Barberio, Assistant Professor, Department of Exercise and Nutrition Science, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCR245732
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Adiposity; Insulin Sensitivity; Impaired Glucose Tolerance; Metabolic Disturbance
Keywords: Metabolism; Feeding; Substrate Oxidation; Metabolic Flexibility; High Fat Diet; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance; Glucose Intolerance | interventions — Diet, High-Fat

STUDY DESIGN:
Intervention Model Description: Non-Randomized Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypercaloric, High Fat Diet (Experimental): For three calendar days participants will be asked to track all foods they eat and beverages they drink (habitual diet) in a mobile application. Following the three days following the habitual diet, participants will consume 165% of their estimated daily energy needs with 65% of those calories coming from fat.
  Interventions: Behavioral: Hypercaloric, High Fat Diet

INTERVENTIONS:
Behavioral: Hypercaloric, High Fat Diet — Participants will select meals from a list of sample breakfast, lunch, and dinner options from grocery stores. Typical intake will be estimated as 160-170% of resting metabolic rate, which will then be multiplied by 1.65 as the target calorie intake for the HFD. Target fat intake will be 65% of the HFD calorie target. To ensure participants will achieve the desired calorie and fat intake, they will also be provided with pre-made nutrient shakes and half-and-half. Participants will supplement their food intake with one to three shakes per day for each of the three days, depending on the fat and calorie content of the foods they select. They will be asked to add half-and-half equally between across the shakes.

SUMMARY:
The purpose of this study is to understand how the body's response after a meal is influenced by insulin and sugar in the blood. The primary question this study seeks to address is what is the effect of reduced insulin sensitivity on postprandial metabolic flexibility to an oral glucose tolerance test. We will recruit 50 adults (ages 20-45; 50% female) who are otherwise healthy (no known clinical diagnosis) into our non-randomized crossover trial to determine the effect of changes in insulin sensitivity on metabolic response to feeding. Insulin sensitivity will be decreased using a three-day high-fat diet (HFD) with extra calories. Whole-body metabolism will be measured during a standard 75-gram oral glucose tolerance test (OGTT). Metabolic response to feeding (e.g. OGTT) will be compared before and after the HFD and compared with the control diet to understand the effect of decreased insulin sensitivity on the metabolic response to feeding. The role of biological sex as a moderator of the effect of increased insulin resistance on postprandial metabolic flexibility will also be investigated

ELIGIBILITY:
Inclusion Criteria:

* Males or Females between the ages of 20 and 45 years
* Body mass index (BMI) of 18.5-29.9 kg/m2
* Low risk for medical complications as determined by physical activity readiness questionnaire (PARQ).
* Low risk for food insecurity via the Hunger Vital Sign screener

Exclusion Criteria:

* Currently taking any antioxidant supplementation, prescription non-steroidal anti- inflammatory drugs, antibiotics, steroids, probiotics, medications for management of cholesterol, diabetes, body weight/obesity, or are undergoing transgender hormone therapy.
* Currently pregnant (verified by urine pregnancy test)
* Any history of disordered eating (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder, etc.) or high risk for disordered eating via validated questionnaire (SCOFF)
* Any history of gastrointestinal diseases (i.e., gastroesophageal reflux disease, irritable bowel syndrome, Celiac disease, Crohn's disease, or lactose intolerance)
* Allergies to wheat or gluten, milk, soy, tree nuts (e.g., almonds, walnuts, pecans), or peanuts.
* Followed a ketogenic diet within the last three months
* Instructed by a medical provided to avoid a high-fat diet due to cardiovascular disease risk.
* Cardiorespiratory fitness (VO2max) greater than the 90th percentile for age and sex

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Postprandial Metabolic Flexibility | 3 Days
  Mean difference respiratory exchange ratio during an oral glucose tolerance test following a high fat diet

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Barberio, PhD, Principal Investigator — George Washington University
Locations (1):
- George Washington University School of Public Health, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No